CLINICAL TRIAL: NCT02772640
Title: The Impact of the Time of Drug Administration on the Effectiveness of Combined Treatment of Hypercholesterolemia With ROSuvastatin and EZEtimibe (ROSEZE) - A Single-center, Crossover, Open-label Study
Brief Title: Effectiveness of Treatment of Hypercholesterolemia With Rosuvastatin and Ezetimibe
Acronym: ROSEZE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Collegium Medicum w Bydgoszczy (Other)
Responsible Party: Principal Investigator, Jacek Kubica, Professor Jacek Kubica MD, PhD., Collegium Medicum w Bydgoszczy
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AMI9
Record Dates: First submitted 2016-03-28; First posted 2016-05-13 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Hypercholesterolemia
Keywords: Hypercholesterolemia; Rosuvastatin; Statin; Ezetimibe; Compliance; Cholesterol; Secondary prevention; Coronary artery disease; Cholesterol absorption inhibitor
MeSH Terms: conditions — Hypercholesterolemia; Patient Compliance; Coronary Artery Disease | interventions — Rosuvastatin Calcium; Ezetimibe

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I: R+E morning->evening (Active Comparator): Rosuvastatin and Ezetimibe morning or evening administration: Rosuvastatin (R) plus Ezetimibe (E) administration in the morning (8:00) for 6 weeks. After 6 weeks - intervention - change of the timing of study drug administration to the evening hours (20:00).
  Interventions: Drug: Rosuvastatin and Ezetimibe morning or evening administration
- ARM II: R+E evening->morning (Active Comparator): Rosuvastatin and Ezetimibe evening or morning administration: Rosuvastatin (R) plus Ezetimibe (E) administration in the evening (20:00) for 6 weeks. After 6 weeks - intervention - change of the timing of study drug administration to the morning hours (8:00).
  Interventions: Drug: Rosuvastatin and Ezetimibe morning or evening administration

INTERVENTIONS:
Drug: Rosuvastatin and Ezetimibe morning or evening administration — Timing of the drug administration:
  morning -> evening evening -> morning
  Other Names: Rosuvastatin, Ezetimibe

SUMMARY:
The aim of the study is to demonstrate, whether the time of day of administration of the study drug (containing rosuvastatin and ezetimibe) has an impact on the effectiveness of lipid-lowering therapy.

DETAILED DESCRIPTION:
The current guidelines recommend statins as drugs of first choice in the treatment of hypercholesterolemia. If the target LDL cholesterol is not achieved, combination of a statin with a cholesterol absorption inhibitor -ezetimibe may be considered.

According to meta-analyzes of studies assessing statins, each 1.0 mmol / L (~ 40 mg / dL) reduction in LDL-C corresponds to a 10% reduction in all-cause mortality and a 20% reduction in the number of deaths from coronary artery disease. Each 1 mmol / L (40 mg / dL) reduction in LDL-C also translates into a 23% and 17% reduction of the risk of major coronary events and stroke, respectively. Similar results concerning the efficacy and safety of lipid-lowering therapy using statins were obtained in meta-analyzes of studies on primary prevention. Statins are a heterogenous group of drugs with respect to their LDL-C reduction power. So far, the most potent statin is rosuvastatin. Despite intensive statin therapy provided, a large group of patients still does not reach therapeutic goals. Statin dose titration seems to be less effective compared with the combined therapy with statin and ezetimibe. The combination of statin with ezetimibe reduces the LDL-C by additional 15-20%.

Tablets comprising both of these drugs (statin and ezetimibe) simplify the drug administration and increase the probability of drug compliance. This may increase the probability for achieving therapeutic goals in hypercholesterolemia treatment.

Taking into account the metabolism of cholesterol and possible drug-drug interactions it is recommended to administer simvastatin in the evening. Rosuvastatin may be administer at any time of the day.

The study is designed as an open-label, single-center, cross-over study evaluating the effectiveness of combined therapy with rosuvastatin and ezetimibe for hypercholesterolemia depending on timing of the day of administration of the study treatment. After enrollment the participants will be allocated into two arms, each receiving rosuvastatin and ezetimibe. The study drug (rosuvastatin with ezetimibe) will be given: 1) in the morning (8:00) for 6 weeks and then in the evening for the next 6 weeks; 2) in the evening (20:00) for the first 6 weeks and then in the morning for the following 6 weeks. The change in total cholesterol and LDL-cholesterol at 6 and 12 weeks of the tested therapy will be measured as the primary outcome of the study. Moreover, other parameters including: HDL-cholesterol, triglycerides, apolipoprotein B (ApoB), ApoAI, nonHDL-cholesterol, sd-LDL-cholesterol, lipoprotein (a), glucose, HBA1c, high sensitivity C reactive protein (hsCRP), ALT, aspartate aminotransferase (AST), creatine kinase (CK ) will be assessed as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Hypercholesterolemia
2. Ineffectiveness of statin monotherapy in the treatment of hypercholesterolemia after at least 6 weeks

Exclusion Criteria:

1. Active liver disease
2. Unexplained persistent increase in serum transaminase levels, including more than 3 times the upper limit of normal activity of one of them
3. Severe renal impairment (creatinine clearance <30 ml / min)
4. Myopathy
5. Concomitant treatment with cyclosporine, gemfibrozil
6. Pregnancy
7. Lactation
8. Women of childbearing age not using effective methods of contraception
9. Symptoms of muscle damage after using statins or fibrates in the past.
10. The activity of creatine kinase> 5 times the upper limit of normal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Change in total cholesterol and LDL-Cholesterol | 6 and 12 weeks
  Change in total cholesterol and LDL-Cholesterol at 6 and 12 weeks of study drug treatment (combination of ezetimibe and rosuvastatin), depending on the time of day of study drug administration

SECONDARY OUTCOMES:
Change in HDL-Cholesterol | 6 and 12 weeks
  Change in HDL-Cholesterol at 6 and 12 weeks of study drug treatment (combination of ezetimibe and rosuvastatin), depending on the time of day of study drug administration
Change in triglycerides | 6 and 12 weeks
  Change in triglycerides at 6 and 12 weeks of study drug treatment (combination of ezetimibe and rosuvastatin), depending on the time of day of study drug administration
Change in apolipoproteins ApoB, APO AI | 6 and 12 weeks
  Change in apolipoproteins ApoB, APO AI at 6 and 12 weeks of study drug treatment (combination of ezetimibe and rosuvastatin), depending on the time of day of study drug administration
Change in non - HDL-Cholesterol | 6 and 12 weeks
  Change in non - HDL-Cholesterol at 6 and 12 weeks of study drug treatment (combination of ezetimibe and rosuvastatin), depending on the time of day of study drug administration
Change in sd-LDL-Cholesterol | 6 and 12 weeks
  Change in sd-LDL-Cholesterol at 6 and 12 weeks of study drug treatment (combination of ezetimibe and rosuvastatin), depending on the time of day of study drug administration
Change in lipoprotein (a) | 6 and 12 weeks
  Change in lipoprotein (a) at 6 and 12 weeks of study drug treatment (combination of ezetimibe and rosuvastatin), depending on the time of day of study drug administration
Assessment of change of glucose concentration | Baseline, 6 and 12 weeks
  Assessment of glucose at baseline and at 6 and 12 weeks of treatment with study drug
Assessment of HbA1c | Baseline, 6 and 12 weeks
  Assessment of HbA1c at baseline and at 6 and 12 weeks of treatment with study drug
Assessment of hsCRP | Baseline, 6 and 12 weeks
  Assessment hsCRP at baseline and at 6 and 12 weeks of treatment with study drug
Assessment of ALT | Baseline, 6 and 12 weeks
  Assessment ALT at baseline and at 6 and 12 weeks of treatment with study drug
Assessment of AST | Baseline, 6 and 12 weeks
  Assessment AST at baseline and at 6 and 12 weeks of treatment with study drug
Assessment of CK | Baseline, 6 and 12 weeks
  Assessment CK at baseline and at 6 and 12 weeks of treatment with study drug
Assessment of plasma fluorescence using stationary and time-resolved spectrofluorimetry | Baseline, 6 and 12 weeks
  Assessment of plasma fluorescence using stationary and time-resolved spectrofluorimetry at baseline, at 6 and 12 weeks of treatment with study drug

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Kubica, MD, PhD, Principal Investigator — Collegium Medicum w Bydgoszczy
Locations (1):
- Cardiology Department, Dr. A. Jurasz University Hospital, Bydgoszcz, Kuyavian-Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Obonska K, Kasprzak M, Sikora J, Obonska E, Racki K, Gozdzikiewicz N, Krintus M, Kubica J. The impact of the time of drug administration on the effectiveness of combined treatment of hypercholesterolemia with Rosuvastatin and Ezetimibe (RosEze): study protocol for a randomized controlled trial. Trials. 2017 Jul 11;18(1):316. doi: 10.1186/s13063-017-2047-8. PMID 28697767
- See also: Study results — https://journals.viamedica.pl/cardiology_journal/article/view/CJ.a2020.0166/52446